CLINICAL TRIAL: NCT02520687
Title: Feasibility Study on the Effects of Dietary Nitrate on Cardiovascular Function in Hypertensive Pregnant Women
Brief Title: Effects of Dietary Nitrate in Hypertensive Pregnant Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manchester (Other)
Responsible Party: Principal Investigator, Dr Jenny Myers, Dr, Manchester University NHS Foundation Trust
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 15136
Record Dates: First submitted 2015-08-05; First posted 2015-08-13 (Estimated); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Hypertension; Pregnancy
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Intervention Model Description: Dietary Nitrate
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dietary nitrate, beetroot juice (Experimental): Once daily 70mL dose of beetroot juice, containing 400mg inorganic nitrate, for 7 consecutive days.
  Interventions: Dietary Supplement: Beetroot juice
- Nitrate-depleted beetroot juice (Placebo Comparator): Once daily 70mL dose of beetroot juice, depleted of nitrate, for 7 consecutive days.
  Interventions: Dietary Supplement: Nitrate-depleted beetroot juice

INTERVENTIONS:
Dietary Supplement: Beetroot juice — 70mls daily for seven days
  Arms: Dietary nitrate, beetroot juice
Dietary Supplement: Nitrate-depleted beetroot juice — 70mls daily for seven days
  Arms: Nitrate-depleted beetroot juice

SUMMARY:
High blood pressure in pregnancy affects around 10% of pregnancies, and is associated with serious adverse outcomes for both mother and baby. Treatment options for the management of high blood pressure in pregnancy are currently limited. Studies in non-pregnant individuals have shown that supplementation with dietary nitrate, using beetroot juice, can significantly lower blood pressure and improve blood flow. This study aims to investigate whether supplementation with dietary nitrate (via beetroot juice) can improve blood pressure regulation in pregnant women with chronic high blood pressure, and will also determine whether this can improve blood flow across the placenta.

ELIGIBILITY:
Inclusion Criteria:

* Women diagnosed with chronic hypertension (systolic blood pressure of 130-144 mmHg and/or diastolic blood pressure of 80-94 mmHg).
* Between 22 - 35+6 weeks gestation

Exclusion Criteria:

* Multi-fetal pregnancy
* Currently taking anti-hypertensive medication
* Pre-existing diabetes (Type 1 or Type 2)
* Lacking ability to consent

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2015-09; Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Change in clinic blood pressure (compared to baseline) between treatment and placebo groups | The outcome will be determined after 7 days treatment (compared to baseline)

SECONDARY OUTCOMES:
Recruitment rates | Across study (18 months)
Uterine artery blood flow (compared to baseline) | The outcome will be determined after 7 days treatment (compared to baseline)
Umbilical artery blood flow (compared to baseline) | The outcome will be determined after 7 days treatment (compared to baseline)
Changes in plasma and salivary nitrate concentrations | The outcome will be determined after 7 days treatment (compared to baseline)
Changes in plasma and salivary nitrite concentrations | The outcome will be determined after 7 days treatment (compared to baseline)

CONTACTS AND LOCATIONS:
Locations (1):
- Maternal and Fetal Health Research Centre, Manchester, United Kingdom